CLINICAL TRIAL: NCT05689541
Title: Development and Refinement of a Parent-mediated Mobile App Intervention for Parents of Children With Autism Spectrum Disorder Participating in an Adapted Horseback Riding Program
Brief Title: Development of a Parent-mediated Mobile App Intervention for Parents of Children With Autism Spectrum Disorder Participating in an Adapted Horseback Riding Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022-0939; EDUC/KINESIOLOGY (Other: UW Madison); 10/6/2022 (Other: Current IRB Application Date)
Record Dates: First submitted 2023-01-09; First posted 2023-01-19 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single group (Other)
  Interventions: Other: Mobile app intervention

INTERVENTIONS:
Other: Mobile app intervention — A mobile-based application will be developed to provide parents with a supplemental curriculum that will include games and activities focusing on motor outcomes. The focus of these games and activities will correspond with the adapted horseback riding program's weekly lesson plan. The mobile app will be created with Glide, which allows us to create a mobile application with basic spreadsheet skills.
  The mobile app will aim to incorporate 10-12 games and activities designed to improve specific motor outcomes. Parents will be instructed to partake in the app-delivered activities with their children daily for at least 30-45 minutes.

SUMMARY:
The purpose of this exploratory sequential mixed methods study is to develop and refine a parent-mediated mobile app intervention focused on improving the motor outcomes of children with autism spectrum disorder (ASD) participating in an adapted horseback riding program.

DETAILED DESCRIPTION:
An exploratory sequential design will be used for the development and refinement of the parent-mediated mobile app. In this three-phase mixed-methods research design, priority will be given to the collection and analysis of the qualitative data in the first phase. Building from the exploratory results of the first phase, the investigator will then conduct a development phase to build the mobile-app intervention. Finally, in the third phase, the investigator will quantitatively assess the acceptability of the newly developed mobile-app intervention.

Qualitative phase:

* Focus group discussions with certified therapeutic riding instructors.
* A semi-structured individual interview will be conducted with parents.

During the focus group with certified therapeutic riding instructors and individual interviews with parents, the previously developed Fit Families app will be presented as a model. The focus group discussions and individual interviews for riding instructors and parents respectively, aim to gain an understanding of the content that will be incorporated into the new parent-mediated mobile app.

The technology acceptance model will guide these interviews and focus group discussions and will be conducted for 45-60 minutes. The technology acceptance model is comprised of four constructs: perceived ease of use, perceived usefulness, attitudes, and actual behaviors. Accordingly, the interview and focus group questions will focus on gaining feedback on aspects such as the user interface, time commitment, different types of games, activities, and homework activities prescribed to children with ASD participating in the adapted horseback riding sessions.

After the initial interviews with the parents and certified therapeutic riding instructors, an approximate time of 6 weeks will be assigned for the development phase. Mid-development interviews with therapeutic riding instructors will guide ongoing development and refine the design/games of the mobile app.

During a group 45-60 minute long training session with the major stakeholders (parents and riding instructors), the fully developed version of the "mobile-app intervention" will be presented. The investigator will train the parents on how to use the mobile app and also answer any questions they might have regarding the usage of the app.

The parents will then be instructed to use the app for two weeks. During this usage period, parents will partake in the games and activities of the app with their children with ASD in their home/community settings.

Similarly, during the training session with the certified therapeutic riding instructors, the mobile app will be presented to understand their perceptions and gain feedback on the first full version of the mobile app intervention.

Quantitative phase:

Upon completion of the 2 weeks implementation period of the newly developed mobile app intervention, parents of children with ASD will be provided with a Qualtrics survey to understand the usability of the app. The parents will be asked to complete a System Usability Scale survey within one week of receiving it.

ELIGIBILITY:
Inclusion Criteria: Parents of children with ASD participating in adapted horseback riding sessions at Three Gaits Inc

* Identify as a parent of a child with ASD ages 6-15
* Have access to a mobile device (mobile phone-iOS or android)
* Be willing to download the mobile app on their device
* Be willing to partake in two focus group interviews each for 45-60 minutes over the summer session
* Be willing to complete the end-of-study survey (approximately 20 minutes)
* English-speaking

Inclusion Criteria: Certified Therapeutic Riding Instructors leading the Adapted Horseback Riding sessions at Three Gaits Inc

* Have a certification (certified therapeutic riding instructor) from the Professional Association of Therapeutic Riding (PATH) Intl.
* Minimum 1 year of experience leading/conducting the adapted horseback riding sessions for children with ASD
* English Speaking

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2023-04-19 (Actual)

PRIMARY OUTCOMES:
Qualitative Exploration of Needs and Perceptions of Participants as measured by Number of Completed Interviews and Focus Group Discussions | up to 2 weeks on study
  The Primary Outcome is to develop a mobile app using qualitative data collected through focus group discussions with therapeutic riding instructors and individual parent interviews; guided by the technology acceptance model. The technology acceptance model is comprised of four constructs: perceived ease of use, perceived usefulness, attitudes, and actual behaviors. Accordingly, the interview and focus group questions will focus on gaining feedback on aspects such as the user interface, time commitment, different types of games, activities, and homework activities prescribed to children with ASD participating in the adapted horseback riding sessions.

SECONDARY OUTCOMES:
Usability of the mobile app as measured by the System Usability Scale Score | 2 weeks post mobile app implementation period (up to 12 weeks on study)
  The System Usability Scale is the most widely used standardized questionnaire for the assessment of the perceived usability of technology/digital tools. Parents use the app for 2 weeks with their children and fill out this survey by rating on a scale of 1 (strongly disagree) to 5 (strongly agree). The participant's scores for each question are converted to a new number, added together and then multiplied by 2.5 to convert the original scores of 0-40 to 0-100. Though the scores are 0-100, these are not percentages and should be considered only in terms of their percentile ranking.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Columna, Principal Investigator — UW-Madison
Locations (1):
- University of Wisconsin- Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No